CLINICAL TRIAL: NCT03576963
Title: A Phase Ib/II Study of Guadecitabine (SGI-110) Plus Nivolumab in Refractory CIMP+ Metastatic Colorectal Cancer
Brief Title: Guadecitabine and Nivolumab in Treating Refractory Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry); Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3C-18-5; NCI-2018-01072 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-18-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-06-21; First posted 2018-07-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Adenocarcinoma; CpG Island Methylator Phenotype; Metastatic Microsatellite Stable Colorectal Carcinoma; Refractory Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — guadecitabine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (guadecitabine, nivolumab) (Experimental): This study consists of an initial dose escalation followed by an expansion cohort. Dose escalation of guadecitabine starts from 30 mg/m^2 given SC on days 1-5 every 28 days in combination with fixed dose of nivolumab at 240 mg given IV on days 8 and 22 every 28 days. Dose escalation will continue until the maximum tolerated dose is reached or all planned doses are administered.
  Interventions: Drug: Guadecitabine; Biological: Nivolumab

INTERVENTIONS:
Drug: Guadecitabine — Given SC
  Other Names: DNMT inhibitor SGI-110; S110; SGI-110
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of guadecitabine when given together with nivolumab and to see how well they work in treating participants with colorectal cancer that does not respond to treatment and has spread to other places in the body. Drugs used in chemotherapy, such as guadecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Giving guadecitabine and nivolumab may work better in treating participants with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability, maximum tolerated dose (MTD)/recommended phase 2 dose (R2PD) of guadecitabine in combination with nivolumab in patients with refractory CpG island methylator phenotype (CIMP+) metastatic colorectal cancer. (Phase Ib Dose Escalation) II. To assess the overall response rate (ORR) in refractory CIMP+ metastatic colorectal cancer patients treated with guadecitabine and nivolumab. (Phase II Expansion)

SECONDARY OBJECTIVES:

I. To determine the incidence of adverse events (AEs) and serious adverse events (SAEs) of guadecitabine combined with nivolumab. (Phase Ib Dose Escalation) II. To assess progression-free (PFS) and overall survival (OS) in refractory CIMP+ metastatic colorectal cancer patients treated with guadecitabine and nivolumab. (Phase II Dose Expansion)

EXPLORATORY OBJECTIVES:

I. Characterize pre and post-treatment morphometric, proteomic and genomic profiles of circulating tumor cells using the high-definition single cell analysis (HD-SCA) platform.

II. Determine associations between circulating cell-free tumor deoxyribonucleic acid (DNA), messenger ribonucleic acid (mRNA) expression, inflammatory T-cell and DNA methylation signatures, with response rate (RR), PFS, OS.

III. Determine associations between tumor PD1/PDL1 expression with RR, PFS, OS.

OUTLINE: This is a phase Ib, dose-escalation study of guadecitabine followed by a phase II study.

Participants receive guadecitabine subcutaneously (SC) on days 1-5 and nivolumab intravenously (IV) over 2 hours on days 8 and 22. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, participants are followed up at 30 days and then every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed microsatellite stable (MSS) metastatic colorectal adenocarcinoma with prior treatment or intolerance to a fluoropyrimidine, oxaliplatin, irinotecan, bevacizumab, and an anti-EGFR agent (in patients with RAS wildtype tumors)
* CIMP+ status: A tumor sample will be classified as CIMP+ if >= 3 of 5 CIMP reactions give a PMR (percent of methylated reference) >= 10, using the MethylLight assay and following CIMP-defining panel - CACNA1G, IGF2, NEUROG1, RUNX3 and SOCS1
* No limit to number of prior lines of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcl
* Serum total bilirubin =< 1.5 upper limit normal (ULN)
* Serum albumin >= 2.5 g/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SPGT]) =< 3 X ULN, unless liver metastases are present or patient has known chronic liver disease, in which case AST and ALT must be =< 5 X ULN
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 5 months after the last dose of study treatment (i.e. 30 days [duration of ovulatory cycle] plus the time required for the investigational drug to undergo approximately five half-lives). Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment (i.e. 90 days [duration of sperm turnover] plus the time required for the investigational drug to undergo approximately five half-lives). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Ability to understand and the willingness to sign a written informed consent
* Patients with treated parenchymal brain metastases are eligible for study participation. Steroids, at stable dose for 2 weeks, not to exceed equivalent of prednisone 10 mg daily dose, are allowed. Anticonvulsants (at stable dose) are allowed. Treatment for brain metastases may be whole-brain radiotherapy, radiosurgery, neurosurgery, or a combination as deemed appropriate by the treating physician. Radiotherapy and stereotactic radiosurgery must be completed at least 28 days prior to randomization

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study (or within 6 weeks for nitrosurea or mitomycin C) or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Any previous treatment with a hypomethylating agent, or with an anti-PD1 or anti-PD-L1 or anti-PD-L2 or anti-CTLA-4 inhibitor, including nivolumab (or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways). Any immunomodulatory agent that is not described above should be cleared by the principal investigator (PI)
* Known hypersensitivity to any of the components of guadecitabine or nivolumab
* Receipt of live attenuated vaccination within 30 days prior to study entry
* History of leptomeningeal carcinomatosis or uncontrolled seizures
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Malignancies other than colorectal adenocarcinoma within 5 years prior to treatment, except for adequately treated carcinoma in situ (e.g. of the cervix), non-melanoma skin cancer, T1a or T1b prostate cancer treated with curative intent at least 1 year prior to study entry with normal prostate specific antigen (PSA), and ductal carcinoma in situ treated surgically with curative intent. Other early stage cancers that have a minimal chance of recurrence (i.e. stage I endometrial cancer, cervical cancer, etc.) may be cleared and should be discussed with the PI
* Renal insufficiency requiring dialysis
* Known positivity for human immunodeficiency virus (HIV)
* Active hepatitis B, hepatitis C
* Surgery (including open biopsy), significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during study treatment
* Active or prior documented autoimmune disease. Subjects with vitiligo, Graves disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn?s disease, ulcerative colitis)
* History of allogeneic organ transplant
* Current or prior use of immunosuppressive medication within 28 days before the first dose of nivolumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Live attenuated vaccines within 30 days of nivolumab dosing (i.e. 30 days prior to the first dose, during treatment with nivolumab and for 30 days post discontinuation of nivolumab. Inactivated vaccines, such as the injectable influenza vaccine, are permitted
* Known history or ongoing diagnosis of pneumonitis
* Known history of previous clinical diagnosis of tuberculosis
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia?s correction
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of guadecitabine when given in combination with nivolumab | Up to 28 days
  MTD defined as the highest dose tested in which none or only one patient experienced dose limiting toxicity (DLT) attributable to the study drug(s), when 6 patients have been treated at that dose and are evaluable for toxicity. DLT defined as toxicity thought to be at least possibly related to study drug(s): Any grade 4 immune related adverse event (irAE); Any > or = grade 3 colitis; Any grade 3 or 4 noninfectious pneumonitis irrespective of duration; Any grade 2 pneumonitis that does not resolve to < or = to grade 1 within 3 days of the initiation of maximal supportive care; Any grade 3 irAE, excluding colitis or pneumonitis, that does not downgrade to grade 2 within 3 days after onset of the event despite optimal medical management including systemic corticosteroids or does not downgrade to < or = grade 1 or baseline within 14 days.
Recommended phase 2 dose (RP2D) of guadecitabine when given in combination with nivolumab | Up to 28 days
  The MTD will be the RP2D, unless other safety considerations intervene. On occasion, the MTD will be expanded to confirm that the doses at the MTD are well tolerated in later courses; if not, a dose lower than the MTD will be selected as the RP2D.

SECONDARY OUTCOMES:
Incidence and severity of adverse events | Up to 1 year
  Will be assessed by Common Terminology Criteria for Adverse Events version 4.03. Will assess frequencies of adverse events (AEs), severe adverse events (SAEs), AEs leading to discontinuation, death, grade 3 and 4 AEs, and grade 3 and 4 laboratory abnormalities occurring up to 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California